CLINICAL TRIAL: NCT00917371
Title: The Effectiveness of Atomoxetine on Brain Imaging, Neuropsychological, and Social Functions in Adults With Attention Deficit/Hyperactivity Disorder
Brief Title: The Effectiveness of Atomoxetine on Brain Imaging, Neuropsychological, and Social Functions in Adults ADHD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200903059M
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2010-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: adults with attention-deficit hyperactivity disorder; atomoxetine; neuropsychological functioning; brain imaging studies
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- atomoxetine group
- methylphenidate group
- psychological counseling group

SUMMARY:
Attention deficit/hyperactivity disorder (ADHD) has been recognized as a common (5-8%), early-onset, long-term impairing, heterogeneous neuropsychiatric disorder with high heritability. Pharmacotherapy (methylphenidate and atomoxetine) has been proved to be the most effective treatment for ADHD. Gau (PI) has done extensive research on ADHD and published 7 SCI papers in ADHD pharmacotherapy. The PI published the first paper in the effectiveness of atomoxetine in improving executive functions among 30 boys with ADHD in the world (International Journal of Neuropsychopharmacology, 2009 Oct 23:1-14. [Epub]). Due to its lifelong impairments up to adulthood, adult ADHD has drawn much more attention in Western studies in the past decade; however, there is lack of such information in Asian population except the PI's three SCI papers on adult ADHD. Because little is known about atomoxetine effect in adults with ADHD except symptoms reduction, this proposal aims to investigate the efficacy of atomoxetine beyond symptoms improvement. The significance of this project is its novelty and research and clinical relevance because there is lack of information regarding long-term effect of atomoxetine on neuropsychological and brain imaging functions on adults with ADHD, a high-prevalent mental disorder with long-term impairment in adults.

DETAILED DESCRIPTION:
Specific Aims:

1. To examine the efficacy of atomoxetine in improving neuropsychological functioning (CANTAB, Time Perception Tasks) and structural (DSI) and functional (resting fMRI) brain connectivity as the primary efficacy endpoints.
2. To examine the efficacy of atomoxetine in reducing ADHD core symptoms and in improving family/social/academic/occupational adjustment and quality of life.

The study design is a randomized open-label, methylphenidate control trial. The sample consists of 60 adults, aged 18-50, with clinical diagnosis of DSM-IV. All participants will be randomly assigned to atomoxetine (n= 30), methylphenidate (n= 15), and clinical visit with psychological counseling (n=15) in a 8-week randomized clinical trial with 3 treatment arms.

The measures included psychiatric interviews (ADHD+SADS), the CGI-ADHD-S, the standardized self-reported questionnaires (the AAQoL, WFIRS-S, and WFIRS-P for social function; ASRS for ADHD symptoms), neuropsychological tests (CANTAB including attention tasks, visual memory, executive functioning, and gambling test; Time Perception Task), and brain imaging (DSI and resting fMRI).

They will be reassessed with safety, ADHD symptoms and social functioning/quality of life at baseline, week 2 (± 5 days), week 4 (± 5 days), and week 8 (± 5 days); neuropsychological tests at baseline, week 4 (± 5 days), and week 8 (± 5 days); and brain imaging studies (DSI and resting-fMRI) at baseline and week 8 (± 5 days). Additionally, blood sample will be collected at baseline for future pharmacogenomic study.

We anticipate that this study will be one of the first to investigate the efficacy of atomoxetine on neuropsychological functioning, and structural and functional brain connectivity in the world. If this research can be carried out, it will be the first project using brain images as assessment tools in a clinical trial among psychiatric patients in psychiatric field in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are (1) that subjects had typical ADHD symptoms before 7 years old which meet the DSM-IV-TR ADHD at childhood and currently based on Gau's clinic diagnosis and the ADHD supplement of the K-SADS for adults; (2) that their Clinical Global Impressions-ADHD-Severity (CGI-ADHD-S) score>4 and psychotropic medication-naïve for the past year; (3) that their IQ greater than 80; and (4) that they consent to this study and they can keep appointments for clinic visits and all tests.

Exclusion Criteria:

These subjects will be excluded from the study if they have any of the following criteria:

* (1) Comorbid with DSM-IV-TR diagnosis of pervasive developmental disorder, schizophrenia, schizoaffective disorder, delusional disorder, other psychotic disorder, organic psychosis, schizotypal personality disorder, bipolar affective disorder, and mental retardation; (2) In the major depressive episode, comorbid with severe anxiety disorders or during substance intoxication or withdrawal at the time of evaluation; (3) With neurodegenerative disorder, epilepsy, involuntary movement disorder, congenital metabolic disorder, brain tumor, history of severe head trauma, and history of craniotomy; (4) A history of alcohol or drug abuse within the past 3 months; (5) The need of psychotropic medications apart from MPH or atomoxetine, including Chinese medicine or health-food supplements that have central nervous system activity; and (6) With visual or hearing impairments, or motor disability which may influence the process of neuropsychological assessment. Subjects will be discontinued from this study in the following circumstances: pregnancy, non-compliance with study drug, an adverse event, subject's request of withdrawal, and loss of follow-up.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will recruit 60 adults, aged 18 to 50, who are diagnosed with ADHD at the PI Gau's Adult ADHD clinic at the Department of Psychiatry, National Taiwan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07-31 (Actual); Study Completion 2011-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lin HY, Gau SS. Atomoxetine Treatment Strengthens an Anti-Correlated Relationship between Functional Brain Networks in Medication-Naive Adults with Attention-Deficit Hyperactivity Disorder: A Randomized Double-Blind Placebo-Controlled Clinical Trial. Int J Neuropsychopharmacol. 2015 Sep 16;19(3):pyv094. doi: 10.1093/ijnp/pyv094. PMID 26377368